CLINICAL TRIAL: NCT04134195
Title: The Effect of Transcranial Direct Current Stimulation on Visual Attention - a Combined MRI and Non-invasive Brain Stimulation Single Session Study
Brief Title: The Effect of Transcranial Direct Current Stimulation on Visual Attention - Single Sessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NV18-04-00256-single
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-09

CONDITIONS: Healthy Aging; Cognitive Change; Cognitive Decline
Keywords: Transcranial direct current stimulation; Healthy seniors; Healthy adults
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real transcranial direct current stimulation (Experimental): Healthy adults and healthy seniors will undergo application of real transcranial direct current stimulation over two distinct brain areas.
  Interventions: Device: Transcranial direct current stimulation
- Sham transcranial direct current stimulation (Experimental): Healthy adults and healthy seniors will undergo application of sham transcranial direct current stimulation over two distinct brain areas.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — 2mA stimulation for 20 minutes

SUMMARY:
Recently, attention has been drawn to non-invasive brain stimulation techniques, such as transcranial direct current stimulation (tDCS), in order to enhance cognitive functions by modifying brain plasticity and use it in different healthy and diseased populations. In the current research, investigator aim to examine the short-term effects of multiple tDCS protocols in healthy adults population on visual attention and identify the neural underpinnings of tDCS-induced behavioral aftereffects using a combined tDCS/ MRI network-based approach.

DETAILED DESCRIPTION:
Investigator will investigate the shor-term effects of active tDCS as compared to a placebo stimulation on visual attention in the healthy seniors. A cross-over, randomized, placebo-controlled design will be used. Single tDCS sessions will be performed in 4 sessions over distinct brain areas with ongoing visual attention training. During the stimulation, investigator will use the visual matching task. MRI protocol consisting of T1 and resting state fMRI sequences will be acquired before and after every stimulation session in order to search for active vs. placebo tDCS-induced changes in brain activation and resting state functional connectivity and to identify neural correlates of behavioral changes.

ELIGIBILITY:
Inclusion Criteria:

* right handed, healthy volunteers in two groups - healthy adults under 40 years, healthy seniors over 50 years

Exclusion Criteria:

* psychiatric disorders, including major depression, major vascular lesions, and other brain pathologies detected by MRI that might present with cognitive decline

  * a cardio pacemaker or any MRI-incompatible metal in the body
  * epilepsy
  * any diagnosed psychiatric disorder
  * alcohol/drug abuse
  * lack of cooperation
  * presence of cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Visual-attention task accuracy | Change from baseline immediately after completion of stimulation protocol
  Task will be presented on a computer and subject will respond by YES-NO buttons. Only if there are no differences in task accuracy, we will measure task reaction times (e.g. due to the roof effect).
Magnetic resonance imaging | Change from baseline immediately after completion of stimulation protocol
  Investigator will record high resolution structural T1-weighted (MPRAGE) images, functional T2* weighted multiband EPI sequences. The total time spent in the scanner will be approximately 40 in every session.

CONTACTS AND LOCATIONS:
Overall Officials: Ľubomira Nováková, Principal Investigator — Ceitec, Masaryk University
Locations (1):
- Ceitec, Masaryk University, Brno, Czechia